CLINICAL TRIAL: NCT01035359
Title: Dorsally Displaced Intraarticular Distal Radius Fractures - Volar Plate or External Fixation. A Prospective Randomized Trial.
Brief Title: Intraarticular Distal Radius Fractures, X-fix or Volar Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sari Ponzer, Professor, MD, Senior consultant orthopaedic surgeon, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRF intra
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Dorsally Displaced Intraarticular Distal Radius Fractures; Age 50 - 74 for Females or 60-74 for Males; Low Energy Trauma
Keywords: radius; fracture; wrist; external; fixation; volar; plate; DASH; PRWE
MeSH Terms: conditions — Fractures, Bone | interventions — External Fixators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- external fixation (Active Comparator): Operation with external fixation and optional addition of k-wire
  Interventions: Procedure: External fixation
- Volar plate (Experimental): Operation with a Synthes volar two column plate (TCP)
  Interventions: Procedure: Volar plate

INTERVENTIONS:
Procedure: External fixation — Bridging external fixation of a distal radius fracture with an optional addition of k-wire(s)
  Other Names: Stryker's Hoffman external fixation
  Arms: external fixation
Procedure: Volar plate — Operation of distal radius fracture with open reduction and fixation with a plate from the volar side of the wrist.
  Other Names: Synthes Two Column Plate (TCP)
  Arms: Volar plate

SUMMARY:
Distal radius fractures are treated surgically if severely displaced. This study aims to investigate the outcome after surgery. The investigators will randomize patients to either external fixation with optional addition of k-wires or open reduction and fixation with a volar plate.

DETAILED DESCRIPTION:
This study has been merged with NCT 01034943 and a new permit has been issued by the Swedish National board on Ethical Permits

ELIGIBILITY:
Inclusion Criteria:

* Female 50-74 years or male 60-74 years
* Dorsally displaced intraarticular distal radius fracture
* Dorsal angulation >20 degrees measured from the plane perpendicular to the radius axis
* Low energy trauma
* Injury <72 hours when diagnosed
* Patient independent of help for ADL

Exclusion Criteria:

* Earlier dysfunction in any wrist
* Other major injuries
* Rheumatoid arthritis or other systemic joint disease
* Dementia or severe psychiatric disease
* Severe medical condition making general anesthesia a major risk

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-08; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is measured by DASH (Disability of the Arm, Shoulder and Hand), which is a self administered questionnaire validated for disease and dysfunction of the upper limb. | 12 months

SECONDARY OUTCOMES:
A secondary outcome is the degree of malalignment on the x-ray of the injured wrist. | 12 months
A secondary outcome of this study is the EQ5D, which is a validated quality-of-life instrument. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm South Hospital Department of Orthopeadic Surgery, Stockholm, Stockholm County, Sweden